CLINICAL TRIAL: NCT01622296
Title: Comparison of Pain of Conventional to Buffered Local Anesthesia During Injection in Pediatric Dental Patients. A Prospective, Double-blind, Randomized, Crossover Study
Brief Title: Comparison of Pain of Conventional to Buffered Local Anesthesia During Injection in Pediatric Dental Patients
Acronym: BufferDent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1107214
Record Dates: First submitted 2012-06-11; First posted 2012-06-19 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Sodium Bicarbonate; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Bicarbonate with Lidocaine (Active Comparator)
  Interventions: Drug: Sodium bicarbonate
- Lidocaine with no buffer (Placebo Comparator)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Sodium bicarbonate — 8.4% neutralizing solution
  Other Names: Sodium Bicarbonate Inj., 8.4% USP Neutralizing Additive Solution (NDC Code 509-100-03)
  Arms: Sodium Bicarbonate with Lidocaine
Drug: Lidocaine — 2% lidocaine with 1:100,000 ppm epinephrine
  Other Names: 2% lidocaine (Brand name: Xylocaine) with 1:100,000 ppm epinephrine, part of the amide family of local anesthetics
  Arms: Lidocaine with no buffer

SUMMARY:
The purpose of this study is to determine the effectiveness of buffered local anesthesia injections to numb the gums and teeth during dental treatment. Adjusting the pH of lidocaine with sodium bicarbonate may reduce the pain of injection for both adults and children. In this study, the investigators will compare two local anesthetic preparations, a buffered anesthetic and the conventionally available anesthetic, for pain upon injection.

Hypothesis: Anesthetic buffered to physiologic pH will result in a less painful injection compared to the acidic alternative used in most dental offices. This can be demonstrated by comparing two local anesthetic preparations, a buffered anesthetic and the conventionally available anesthetic, for pain upon injection.

DETAILED DESCRIPTION:
Local anesthesia is an essential procedure in the comprehensive treatment of pediatric patients. In the treatment of subjects with dental disease and infection, local anesthesia is commonly required when performing operative procedures. The use of local anesthesia serves two main purposes: (i) enables the patient to remain free of discomfort during the sometimes painful procedure and (ii) permits the practitioner to complete the procedure without fear of hurting the patient which might otherwise impede the practitioner's ability to provide comprehensive care. However, patients are often fearful of local anesthesia because traditional preparations of local anesthesia are acidic and can be painful. Thus, an important advance in the areas of subject management and pain control during operative procedures would be a preparation of local anesthesia that significantly reduced the pain upon injection. A 2010 Cochrane Review found that adjusting the pH of lidocaine with sodium bicarbonate reduced the pain of injection for both adults and children. In this study, we will compare two local anesthetic preparations, a buffered anesthetic and the conventionally available anesthetic, for pain upon injection.

The study will test a local anesthetic buffering system, the Onset system, an FDA Class 1 compounding device manufactured by Onpharma Inc. It is a simple and portable local anesthesia buffering system that compounds anesthetic solution and 8.4% sodium bicarbonate neutralizing additive solution in a precise manner that brings the anesthetic solution up to human physiologic pH. Commercially available local anesthetics have a low pH to allow for prolonged shelf life, and to keep the anesthetic molecules in solution. The combination of a buffering sodium bicarbonate agent and local anesthetic has been reported to result in pain-free injections for both adults and children. The neutralizing additive solution is a sterile, nonpyrogenic, solution of sodium bicarbonate (NaHCO3) in water. pH is adjusted with carbon dioxide. Sodium Bicarbonate Inj., 8.4% USP Neutralizing Additive Solution (NDC Code 509-100-03) and Lidocaine w/ Epinephrine are compatible. Sodium bicarbonate is used in medicine and dentistry as regularly as saline, and pre-dates the FDA. It is commercially available and currently being used by health professionals in the U.S.A.

The local anesthetic used in the study will be 2% lidocaine with 1:100,000 ppm epinephrine, part of the amide family of local anesthetics. It has been widely used in dentistry and medicine and has long-standing proven records of safety.

ELIGIBILITY:
Inclusion Criteria:

* Give written, informed consent (both the subject and the legal guardian)
* Be 9-12 years of age
* Be able to comprehend the visual analog scale (instructions given to ascertain this)
* Be able to comprehend the verbal rating scale (instructions given to ascertain this)
* In the opinion of the investigator, be a subject who can be expected to comply with the protocol
* Present moderate mandibular dental disease bilaterally
* Have 4 to 7 natural teeth (with at least one posterior tooth) present in each mandibular quadrant with moderate dental disease on at least one tooth
* Be willing to attend the clinic for 3 or more appointments

Exclusion Criteria:

* Antibiotic premedication requirement
* A history of allergy, sensitivity, or any other form of adverse reactions to local anesthetics of the amide type, or epinephrine
* A history of specific systemic illness that would preclude administration of a local anesthetic or vasoconstrictor (epinephrine) (e.g. liver , renal, cardiovascular diseases, blood dyscrasias, psychiatric disorders, etc.)
* A history of systemic illness that would interfere with healing response (e.g. liver disease, blood dyscrasias, uncontrolled diabetes, etc.)
* Current systemic medication that interferes with healing response
* Current systemic medication which contraindicates the use of local anesthetics or epinephrine
* Pregnant or lactating females (contradicts the use of local anesthetic in non-emergency type dental procedures)
* Current alcohol or drug abuse
* Received an anesthetic, analgesic or sedative within 24 hours prior to the therapy appointments
* Acute infections or conditions in the oral cavity requiring immediate treatment
* Participation in a clinical study of an investigational drug within the previous 4 weeks
* Previous enrollment in the present study

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Tavana, DDS, Principal Investigator — University of Caifornia, San Francisco; Peter Loomer, DDS, PhD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Milgrom P, Coldwell SE, Getz T, Weinstein P, Ramsay DS. Four dimensions of fear of dental injections. J Am Dent Assoc. 1997 Jun;128(6):756-66. doi: 10.14219/jada.archive.1997.0301. PMID 9188235
- [Background] Cepeda MS, Tzortzopoulou A, Thackrey M, Hudcova J, Arora Gandhi P, Schumann R. Adjusting the pH of lidocaine for reducing pain on injection. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD006581. doi: 10.1002/14651858.CD006581.pub2. PMID 21154371
- [Background] von Baeyer CL. Children's self-report of pain intensity: what we know, where we are headed. Pain Res Manag. 2009 Jan-Feb;14(1):39-45. doi: 10.1155/2009/259759. PMID 19262915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 healthy pediatric volunteers were recruited at one U.S. clinical site. All participants completed both study interventions.
Groups:
- Lidocaine First, Then Buffered Lidocaine: lidocaine 2% with 1:100,000 epinephrine followed by buffered lidocaine 2% with 1:100,000 epinephrine. Two treatment visits were required to complete bilateral dental operative restorations. At each visit, local anesthetic was delivered to the right or left side of the dentition using one of the two anesthetic types. The second injection/treatment appointment was at least 1 week after the first treatment.
- Buffered Lidocaine First, Then Lidocaine: buffered lidocaine 2% with 1:100,000 epinephrine followed by lidocaine 2% with 1:100,000 epinephrine. Two treatment visits were required to complete bilateral dental operative restorations. At each visit, local anesthetic was delivered to the right or left side of the dentition using one of the two anesthetic types. The second injection/treatment appointment was at least 1 week after the first treatment.
Period: First Intervention
Arm/Group | Lidocaine First, Then Buffered Lidocaine | Buffered Lidocaine First, Then Lidocaine
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Period of at Least 1 Week
Arm/Group | Lidocaine First, Then Buffered Lidocaine | Buffered Lidocaine First, Then Lidocaine
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Lidocaine First, Then Buffered Lidocaine | Buffered Lidocaine First, Then Lidocaine
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: per protocol
Groups:
- Crossover Lidocaine/Buffered Lidocaine: lidocaine 2% with 1:100,000 epinephrine followed by buffered lidocaine 2% with 1:100,000 epinephrine or buffered lidocaine 2% with 1:100,000 epinephrine followed by lidocaine 2% with 1:100,000 epinephrine
Arm/Group | Crossover Lidocaine/Buffered Lidocaine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 10 [9 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Participant Pain Experience After Administration of Local Anesthesia to Numb the Gums and Teeth During Dental Treatment
Description: Two treatment visits were required for bilateral, mandibular dental operative restorations. At each visit, local anesthetic was delivered to the right or left side of the dentition using one of the two anesthetic types. The administering operator stepped out of the room after each injection was completed, and the participant was asked by a trained research assistant to record a visual analog scale (VAS) pain score. The VAS was used to assess pain sensitivity, and utilizes a 100mm horizontal line, with scores ranging from 0 ("no pain") to 100 ("pain as bad as it can be").
Time Frame: immediately after anesthetic injection
Population: per protocol, in a crossover fashion, each participant received buffered lidocaine at one treatment visit and lidocaine at one treatment visit, in randomly assigned sequence.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Buffered Lidocaine: 2% buffered lidocaine with 1:100,000 ppm epinephrine
Arm/Group | Lidocaine | Buffered Lidocaine
Number analyzed (Participants) | 20 | 20
units on a scale
  Pain on inferior alveolar nerve block | 43 (6) | 33.1 (5.5)
  Pain on long buccal nerve block | 7.3 (1.9) | 9.8 (3.9)
Statistical Analysis 1: Comparison: Lidocaine vs Buffered Lidocaine; Inferior Alveolar nerve injection - H(0): Lidocaine VAS score = Buffered Lidocaine VAS score. Based on data from medial trials of buffered anesthetic, a power calculation for sample size indicated that 20 subjects would provide a 90% change of detecting an effect size of 0.83 (a change of 0.83 standard deviations); Test type: Superiority or Other; p = 0.23, t-test, 2 sided — Significant at p<0.05
Statistical Analysis 2: Comparison: Lidocaine vs Buffered Lidocaine; Long buccal nerve injection - H(0): Lidocaine VAS score = Buffered Lidocaine VAS score. Based on data from medial trials of buffered anesthetic, a power calculation for sample size indicated that 20 subjects would provide a 90% change of detecting an effect size of 0.83 (a change of 0.83 standard deviations); Test type: Superiority or Other; p = 0.57, t-test, 2 sided — Significant at p<0.05

ADVERSE EVENTS:
Time Frame: up to 48 hours after treatment procedures
Description: Participants were contacted by telephone within 48 hours and asked standardized follow-up questions to determine if there were any adverse reactions: 1. Have you had any health problems since you left the dental clinic?, 2. Have you had any soreness in your mouth since you left the dental clinic?, 2.a. If yes, is the soreness at the injection site?
Arm/Group | Crossover Lidocaine/Buffered Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
The variation of VAS scores was found to be larger than that used in the sample size calculation; thus, the study was underpowered to reach statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes